CLINICAL TRIAL: NCT02411136
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 623 Following Multi-dose Administration in Subjects With Systemic Lupus Erythematosus
Brief Title: A Study to Examine the Safety, Pharmacokinetics and Pharmacodynamics of AMG 623 in Subjects With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20040250
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMG 623 (Experimental): Multiple doses of AMG 623 administered as subcutaneous and intravenous doses
  Interventions: Drug: AMG 623
- Placebo (Placebo Comparator): Multiple doses of AMG 623 administered as subcutaneous and intravenous doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 623 — Multiple doses of AMG 623 administered as subcutaneous and intravenous doses
  Arms: AMG 623
Drug: Placebo — Multiple doses of AMG 623 administered as subcutaneous and intravenous doses
  Arms: Placebo

SUMMARY:
This study is to evaluate the safety of AMG 623 in subjects with systemic lupus erythematosus. All subjects will receive 4 weekly doses of study drug over a 3 week period, and then will be followed for an additional 28 weeks, for total study duration of 31 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 65 years old
* Diagnosis of SLE
* Stable disease; defined as no change in SLE therapy within the previous 30 days. Up to 5 mg/day incremental changes of prednisone therapy is allowed during the 30 days prior to randomization
* SLE disease duration of at least 1 year, as diagnosed by a physician

Exclusion Criteria:

* Current renal disease
* Signs or symptoms of viral or bacterial infection within 30 days of enrollment
* Any disorder (including psychiatric), condition or clinically significant disease (other than a diagnosis of SLE) that would interfere the study evaluation, completion and/or procedures per the investigator's discretion
* Administration of more than 10 mg/day prednison (or equivalent) in the 30 days prior to randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-05; Primary Completion 2007-08 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | up to 31 weeks
Incidence of abnormal clinically significant vital signs | up to 31 weeks
Incidence of abnormal clinically significant chemistry, hematology and urinalysis test results | up to 31 weeks
Incidence of abnormal clinically significant ECG results | up to 31 weeks

SECONDARY OUTCOMES:
Pharmacokinetics profile of AMG 623 including Tmax, AUClast and Cmax | up to 31 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Stohl W, Merrill JT, Looney RJ, Buyon J, Wallace DJ, Weisman MH, Ginzler EM, Cooke B, Holloway D, Kaliyaperumal A, Kuchimanchi KR, Cheah TC, Rasmussen E, Ferbas J, Belouski SS, Tsuji W, Zack DJ. Treatment of systemic lupus erythematosus patients with the BAFF antagonist "peptibody" blisibimod (AMG 623/A-623): results from randomized, double-blind phase 1a and phase 1b trials. Arthritis Res Ther. 2015 Aug 20;17(1):215. doi: 10.1186/s13075-015-0741-z. PMID 26290435
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com